CLINICAL TRIAL: NCT00012662
Title: Disease Management and Educational Intervention Outcomes in High-Risk Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DII 99-188
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Diabetes Mellitus Self Management Education; Hyperglycemic Control; High Risk Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Diabetes Self Management Education

INTERVENTIONS:
Behavioral: Diabetes Self Management Education

SUMMARY:
Social, medical and economic burdens of diabetes care result from microvascular, macrovascular and neurological complications. Sustained reduction in hyperglycemia can reduce the incidence of these complications by as much as 50 percent. Studies have demonstrated improved glycemic control with nurse case-management or educational care models. However, none have controlled for their independent contributions, intervened with advanced practice nurses (APN), or targeted highest risk individuals.

DETAILED DESCRIPTION:
Background:

Social, medical and economic burdens of diabetes care result from microvascular, macrovascular and neurological complications. Sustained reduction in hyperglycemia can reduce the incidence of these complications by as much as 50 percent. Studies have demonstrated improved glycemic control with nurse case-management or educational care models. However, none have controlled for their independent contributions, intervened with advanced practice nurses (APN), or targeted highest risk individuals.

Objectives:

The objective of this project is to examine whether interventions of diabetes self-management education programs with or without APN case managers improve outcomes and are cost effective.

Methods:

Patients were randomly assigned to one of four groups: 1) Disease-management and diabetes education; 2) Disease-management alone; 3) Diabetes education alone; and 4) Routine Care. Veterans receiving primary care in VISN-5 and meeting high-risk criteria (HbA1c � 9.0%) were screened for inclusion. Patient outcome measures were collected at baseline, three months and twelve months. These included: Quality of Life (QOL), HgbAlc levels, and incidence of diabetes-related hospitalizations/ER visits. In addition, patient-level intervention costs, health care use and costs were examined. ANOVA comparisons were used to test hypotheses.

Status:

Recruitment is over and final analyses are underway.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes HbA1C. 9.0%, consistent diabetes tx over last 3 months.

Exclusion Criteria:

Homelessness-not able to be consistently contacted; Dementia, Planned Movement from area; Unstable angina, Myocardial Infarction in past 3 months; Stroke; Two or more seizures in last 3 months; document alcoholism or drug abuse; Pregnant or planning to become pregnant in next 12 months; Severe immunodeficiency or cirrhosis of the liver; Type 1 diabetes; blind individuals; psychosis; pancreatitis with secondary diabetes; Renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce P. Hamilton, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Atlanta, Kansas, United States

REFERENCES:
- [Result] Bradham DD, Mangan M, Warrick A, Geiger-Brown J, Reiner JI, Saunders HJ. Linking innovative nursing practice to health services research. Nurs Clin North Am. 2000 Jun;35(2):557-68. PMID 10873268